CLINICAL TRIAL: NCT06812273
Title: Mediators and Moderators of Auditory Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Oregon Health and Science University (Other); University of California, Riverside (Other)
Responsible Party: Principal Investigator, Aaron Seitz, Professor of Psychology, Game Design, and Physical Therapy, Movement and Rehabilitation Services, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22066
Record Dates: First submitted 2025-01-21; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Hearing Handicap
Keywords: audition; auditory training; cognition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- STM Training (Experimental)
  Interventions: Behavioral: STM Training
- Speech Training (Experimental)
  Interventions: Behavioral: Speech Training
- Mixed Training (Experimental)
  Interventions: Behavioral: Mixed Training
- Gamified Training (Experimental)
  Interventions: Behavioral: Gamified Training
- Foraging Training (Experimental)
  Interventions: Behavioral: Foraging Training
- Business As Usual (No Intervention)

INTERVENTIONS:
Behavioral: STM Training — This condition consists of an up/down spectral-temporal modulations (STM) presented both in quiet and with competing background noise
  Arms: STM Training
Behavioral: Speech Training — Participants will train on the identification of three sets of speech stimuli of increasing linguistic complexity: individual phonemes (vowels), spondaic words, and matrix sentences.
  Arms: Speech Training
Behavioral: Mixed Training — This condition involves both the STM and the speech training, described above, and an additional module training localization.
  Arms: Mixed Training
Behavioral: Gamified Training — This uses auditory training within a game experience where players control a game avatar (the "wisp") that appears to fly through a landscape. Players were asked to help the wisp avoid obstacles or choose from among options based on a variety of sound cues.
  Arms: Gamified Training
Behavioral: Foraging Training — This adds a component to the game where participants navigate the wisp to the location on the screen that relates to the target stimulus. The concept here is that searching for targets with manual movements, ecologically stimulates sensori-motor loops where the actions of the participants generates the auditory stimuli that are heard.
  Arms: Foraging Training

SUMMARY:
The goal of this clinical trial is to learn how Auditory Training (AT) may help people better understand speech in noisy environments. As people get older, it becomes harder for them to hear speech clearly when there is background noise. This can be frustrating, and it can affect their independence and quality of life. AT is often used to support people with and without hearing loss, especially when a person is not a good candidate for a hearing aid or when amplification from a hearing aid does not improve performance.

The investigators want to gather reliable data to understand how AT works and what affects its success.

The main questions the trial aims to answer are:

* How do different types of sounds influence the effectiveness of auditory training?
* Which auditory training approaches are most successful in improving speech understanding?
* How do personal traits impact the results of auditory training?

The investigators will study a large and diverse group of 1,260 participants, including both young and older adults, to evaluate various auditory training approaches.

You will:

* Take part in auditory training sessions that include different types of auditory tasks.
* Complete tests that measure how well they understand speech in both quiet and noisy settings.
* Complete surveys on personal data like demographics, hearing challenges and other factors to help researchers understand what might influence training results.

The investigators will measure and compare the results of these approaches to find out which ones are most effective. This could help people who are at risk of cognitive decline, like those at risk for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 and 60-85 years of age.
* No self-reported auditory difficulties and normal or near-normal hearing sensitivity as measured by SRTs.
* Older adults aged 50-85 should have no more than typical hearing loss for their age and no evidence of dementia.
* Fluent in English and/or Spanish

Exclusion Criteria:

* Abnormal vision or hearing prohibitive of training
* History of seizures, focal brain lesion, or head injury with loss of consciousness
* Physical handicap (motor or perceptual) that would impede training procedures
* Medical illness requiring treatment during the study timeline
* Social, educational or economic hardship prohibitive to training schedule
* Concurrent enrollment in other cognitive training studies
* History of major psychiatric illness, including psychosis, bipolar disorder, depression, alcohol or substance abuse, recent bereavement
* Plans to travel out of the area for more than 1 week during the intervention period
* Residence too far from the testing site, which would prevent attending the testing sessions (> 60 miles)
* Not being proficient enough in English or Spanish that would prevent following and understanding all instructions and completing all testing sessions

Additional exclusion criteria for older adults:

* Diagnosis of dementia or other neurological disease, including mild cognitive impairment (MCI)
* Telephone-Montreal Cognitive Assessment (t-MoCA) score of 16 or less or Montreal Cognitive AssessmentMoCA) score of 20 or less

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Digits-in-Noise (DIN) Task | Pre-test (day 3), mid-test (day 20), post-test (day 36), follow-up (day 66)
  The DIN tests the ability to identify a series of digits in varying levels of background noise.
Spatial Release From Masking (SRM) | Pre-test (day 3), mid-test (day 20), post-test (day 36), follow-up (day 66)
  Tests the ability to identify a target talker in the presence of competing speech signals that are either colocated or spatially separated from the target.
Dichotic Sentence Identification (DSI) | Pre-test (day 3), mid-test (day 20), post-test (day 36), follow-up (day 66)
  The DSI test simultaneously presents two nonsense sentences, one to each ear. Participants indicate two sentences heard from a list of 10 alternatives.

SECONDARY OUTCOMES:
Revised Hearing Handicap Inventory (RHHI) | Pre-test (day 3), mid-test (day 20), post-test (day 36), follow-up (day 66)
  The Revised Hearing Handicap Inventory (RHHI) is a self-assessment questionnaire designed to evaluate the perceived social and emotional effects of hearing loss on an individual's daily life.
Auditory Visual Divided Attention Test (AVDAT) | Pretest (day 3), post-test (day 36), follow-up (day 66)
  Auditory Visual Divided Attention Test (AVDAT) is a test of working memory that compares conditions when attention is to just a single modality (auditory or visual) or divided across modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Seitz, PhD, Principal Investigator — Northeastern University; Tess Koerner, PhD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - University of California, Riverside, Riverside, California
  - Northeastern University, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria.